CLINICAL TRIAL: NCT02722265
Title: Open-label, Multicenter, Interventional, Dose Titration Study to Assess the Long-term Study of CS-3150 2.5mg and 5mg Alone as Monotherapy or in Combination With Other Antihypertensive Drug in Japanese Patients With Essential Hypertension
Brief Title: Long-term Study of CS-3150 as Monotherapy or in Combination With Other Antihypertensive Drug in Japanese Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3150-A-J302
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; Long-term treatment; Mineralocorticoid receptor antagonist
MeSH Terms: conditions — Essential Hypertension | interventions — esaxerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS-3150 (Experimental): CS-3150 2.5mg to 5mg, orally, once daily for 28 or 52 weeks
  Interventions: Drug: CS-3150

INTERVENTIONS:
Drug: CS-3150 — CS-3150 2.5mg to 5mg, orally, once daily for 28 or 52 weeks

SUMMARY:
To examine antihypertensive effect, pharmacodynamics, and safety of long-term administration of CS-3150 as monotherapy and in combination with calcium channel blocker or renin-angiotensin system inhibitor in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20 years or older at informed consent
* Subjects with essential hypertension, who do not receive any antihypertensive drugs or receive calcium channel blocker, angiotensin converting enzyme ACE inhibitor, or angiotensin-II receptor blockade ARB during run-in period (Sitting systolic blood pressure SBP ≥ 140 mmHg and < 180 mmHg, Sitting diastolic blood pressure DBP ≥ 90 mmHg and < 110 mmHg, and mean 24hr SBP ≥ 130 and DBP ≥ 80 mmHg)

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* Diabetes mellitus with albuminuria
* Serum potassium level < 3.5 or ≥ 5.1 mEq/L (≥ 4.8 mEq/L if receive ACE inhibitor, or ARB)
* Reversed day-night life cycle including overnight workers
* estimated glomerular filtration rate eGFR < 60 mL/min/1.73 m^2.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07-08 (Actual); Study Completion 2017-07-08 (Actual)

PRIMARY OUTCOMES:
change from baseline in sitting systolic and diastolic blood pressure | week 0 (baseline) to end of weeks 12, 28, and 52

SECONDARY OUTCOMES:
Change from baseline in 24-hr ambulatory blood pressure monitoring (ABPM) | week 0 (baseline) to end of weeks 12, 28, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo Co., Ltd.
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Ichikawa S, Tsutsumi J, Sugimoto K, Yamakawa S. Antihypertensive Effect of Long-Term Monotherapy with Esaxerenone in Patients with Essential Hypertension: Relationship Between Baseline Urinary Sodium Excretion and Its Antihypertensive Effect. Adv Ther. 2022 Oct;39(10):4779-4791. doi: 10.1007/s12325-022-02282-3. Epub 2022 Aug 17. PMID 35976603